CLINICAL TRIAL: NCT02754895
Title: Positive Psychology for Acute Coronary Syndrome Patients: a Factorial Design Study
Brief Title: Positive Psychology for ACS Patients: a Factorial Design Study
Acronym: PEACEIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director of Inpatient Psychiatric Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P001756; 4R01HL113272-04 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; health behavior; factorial design; positive psychology
MeSH Terms: conditions — Acute Coronary Syndrome; Health Behavior | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- PP-weekly (Experimental): Participants will receive the positive psychology intervention and will be asked to complete a PP exercise once per week.
  Interventions: Other: Positive Psychology (PP)
- PP-daily (Experimental): Participants will receive the positive psychology intervention and will be asked to complete a PP exercise once per day.
  Interventions: Other: Positive Psychology (PP)
- Shortened PP-weekly plus MI (Experimental): Participants will receive a shortened version of the positive psychology intervention in addition to motivational interviewing and will be asked to complete a PP exercise once per week.
  Interventions: Other: Positive Psychology (PP); Other: Motivational Interviewing (MI)
- Shortened PP-daily plus MI (Experimental): Participants will receive a shortened version of the positive psychology intervention in addition to motivational interviewing and will be asked to complete a PP exercise once per day.
  Interventions: Other: Positive Psychology (PP); Other: Motivational Interviewing (MI)
- PP-weekly with boosters (Experimental): Participants will receive the positive psychology intervention and will be asked to complete a PP exercise once per week. Participants will also receive three "booster" phone calls following the completion of the 8 week intervention.
  Interventions: Other: Positive Psychology (PP)
- PP-daily with boosters (Experimental): Participants will receive the positive psychology intervention and will be asked to complete a PP exercise once per day. Participants will also receive three "booster" phone calls following the completion of the 8 week intervention.
  Interventions: Other: Positive Psychology (PP)
- Shortened PP-weekly plus MI + boosters (Experimental): Participants will receive a shortened version of the positive psychology intervention in addition to motivational interviewing and will be asked to complete a PP exercise once per week. Participants will also receive three additional "booster" phone calls following the completion of the 8 week intervention.
  Interventions: Other: Positive Psychology (PP); Other: Motivational Interviewing (MI)
- Shortened PP-daily plus MI with boosters (Experimental): Participants will receive a shortened version of the positive psychology intervention in addition to motivational interviewing and will be asked to complete a PP exercise once per day. Participants will also receive three additional "booster" phone calls following the completion of the 8 week intervention.
  Interventions: Other: Positive Psychology (PP); Other: Motivational Interviewing (MI)

INTERVENTIONS:
Other: Positive Psychology (PP) — Positive psychology (PP) interventions aim to improve the frequency and intensity of positive emotional experiences. This positive psychology intervention focuses on targeted activities in several domains, including altruism (e.g., performing acts of kindness), gratitude (e.g., systematically recalling positive life events), using one's personal strengths in a deliberate manner, and optimism (e.g., thinking about past successes and applying these skills to the future).
Other: Motivational Interviewing (MI) — MI is a goal-oriented, patient-centered approach to helping patients resolve their ambivalence to change their health behaviors.
  Each session follows the same structure. Study trainers will: (a) ask participants about their health goals, (b) advise them about current health guidelines and/or refer them to their treatment team, (c) assess readiness to set a goal by identifying how important participants feel the goal is, how confident participants are about making a change, and what the participants' pros and cons for making a change, (d) assist participants in clarifying their goals and problem-solving barriers to reaching those goals, and (e) arrange for the next session by summarizing the participant's plan and scheduling the next session.
  Arms: Shortened PP-daily plus MI; Shortened PP-daily plus MI with boosters; Shortened PP-weekly plus MI; Shortened PP-weekly plus MI + boosters

SUMMARY:
This trial is part of a multi-phase study to develop and test positive psychology (PP) interventions in patients hospitalized for an acute coronary syndrome (ACS).Using a factorial design, the investigators will: (a) assess the optimal frequency of exercise completion, (b) determine the utility of 'booster sessions' after an initial 8-week intervention, and (c) determine the relative merits of utilizing PP exercises alone versus an intervention combining PP with motivational interviewing (MI).

DETAILED DESCRIPTION:
The investigators have completed the intervention development and pilot phases (PEACE and PEACEII), and are now aiming to optimize our PP intervention for the target population prior to testing it in a randomized, controlled trial.

The investigators will recruit patients from MGH and Brigham and Women's Hospital (BWH) inpatient units who are admitted with a primary cardiac diagnosis of ACS. Following the completion of baseline outcome measures, participants will be randomized to one of eight treatment conditions. All participants will complete PP exercises at least weekly and will speak with a study trainer weekly for eight weeks. Those receiving the PP-only intervention (conditions 1, 2, 5, 6) will speak to a study trainer for 30 minutes each week. Participants in Conditions 3, 4, 7, and 8 will be enrolled in a combined PP plus motivational interviewing (MI)/goal setting program. Accordingly, their weekly phone sessions will focus on the PP program for 15 minutes, then the MI/goal setting program for an additional 15 minutes. These calls will be recorded, and a percentage of calls will be reviewed to ensure that the PP and MI/goal setting portions of the intervention are being delivered as described in the protocol and trainer manual. Half of the participants (conditions 1, 3, 5, 7) will be instructed to perform the PP exercises once per week while the other half (conditions 2, 4, 6, 8) will be asked to perform them once daily. Finally, half of the participants (those in conditions 5-8) will receive three additional 'booster' phone sessions during weeks 10, 12, and 14. These sessions will focus on integrating PP-related skills into daily life. For participants in the PP+MI condition, booster sessions also will focus on maintaining the health behavior changes that they made during the main portion of the study.

The PP exercises used in this study were selected based on their superior performance in our pre-pilot research and others' work: Gratitude for Positive Events (Week 1), Using personal strengths (Week 2), Gratitude letter/Expressions of Gratitude (Week 3), Capitalizing on Positive Events (Week 4), Remembering past success/Remembering daily successes (Week 5), Enjoyable and meaningful activities (Week 6), Humor in everyday life (Week 7), and Performing acts of kindness & Next Steps (Week 8). Participants in conditions 5-8 will have three additional bi-weekly "maintaining your gains" sessions (week 10, 12, and 14) in order to identify favorite exercises, explore the skills derived from doing the exercises, and learn how to integrate the exercises in their daily lives.

For the MI/goal setting portion of the intervention, each session follows the same structure. Study trainers will: (a) ask participants about their health goals, (b) advise them about current health guidelines and/or refer them to their treatment team, (c) assess readiness to set a goal by identifying how important participants feel the goal is, how confident participants are about making a change, and what the participants' pros and cons are for making a change, (d) assist participants in clarifying their goals and problem-solving barriers to reaching those goals, and (e) arrange for the next session by summarizing the participant's plan and scheduling the next session. The structure of the sessions will follow the PP structure according to each condition.

At Weeks 8 and 16, a member of the study staff will call participants to repeat the self-report questionnaires that were administered at baseline. Furthermore, at Weeks 8 and 16, participants will wear an ActiGraph step counter for 10 days as a measure of physical activity. At 3 and 6 months post enrollment, a research coordinator will call participants to ask some brief questions concerning their health, well-being, adherence to health behaviors, and the application of positive psychology and motivational interviewing skills in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to MGH or BWH inpatient units
* Diagnosis of acute coronary syndrome (using established criteria for myocardial infarction or unstable angina; confirmed via medical record and/or patient's treatment team)
* Age 18 or older
* Suboptimal adherence on MOS-SAS: Score < 15 OR Score = 15 with physical activity < 6

Exclusion Criteria:

* Cognitive deficits, assessed with 6-item screen
* Inability to participate in physical activity
* Medical conditions precluding interviews or likely to lead to death within 6 months
* Inability to read/write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Physical activity | 16 weeks (primary outcome for all analyses)
  To assess which components of the intervention (daily vs. weekly exercise completion, booster vs. no booster sessions, PP only vs. PP + MI) are associated with the greatest physical activity measured by the Actigraph accelerometer (steps) at 16 weeks.

SECONDARY OUTCOMES:
Change in adherence to health behaviors, main secondary outcome | Baseline, 8 week, 16 week
  Measured by the three items from the Medical Outcomes Study-Specific Adherence Scale (MOS SAS)
Change in self-report adherence to physical activity | Baseline, 8 week, 16 week
  Measured by one item from the Medical Outcomes Study-Specific Adherence Scale (MOS SAS) which specifically asks about physical activity.
Change in positive affect | Baseline, 8 week, 16 week
  Measured by the Positive and Negative Affect Schedule (PANAS)
Change in optimism | Baseline, 8 week, 16 week
  Measured by the Life Orientation Test-Revised (LOT-R)
Change in anxiety | Baseline, 8 week, 16 week
  Measured by the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
Change in depression | Baseline, 8 week, 16 week
  Measured by the depression subscale of the Hospital Anxiety and Depression Scale (HADS)
Change in physical function | Baseline, 8 week, 16 week
  Measured by the Duke Activity Status Index (DASI)
Change in health-related quality of life (HRQoL) | Baseline, 8 week, 16 week
  Measured by the Short Form 12 (SF-12)
Change in medication adherence | Baseline, 8 week, 16 week
  Measured by self-report
Change in dietary adherence | Baseline, 8 week, 16 week
  Measured by the MEDFICTS scale, a National Cholesterol Education Program-developed scale inquiring about saturated fat

OTHER OUTCOMES:
Feasibility of the intervention | 16 weeks
  Measured using rates of session completion (i.e., completion of both the prior week's PP activity and the session call) and completion of study follow-up assessments (including self-report phone assessments, accelerometer use, and use of the electronic pillcaps).
Acceptability of the intervention | 16 weeks
  Measured by weekly 0-10 ratings of each PP exercise. Positive affect and optimism are rated immediately prior to completing the assigned PP exercise for that week and then immediately following completion of the exercise. Also, the participants provide post-exercise ratings of the exercise's ease of completion and utility.
Overall effect of intervention | 16 weeks
  Measured by pre-post changes in self-reported adherence, depressive symptoms, anxiety, optimism, and positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duque L, Brown L, Celano CM, Healy B, Huffman JC. Is it better to cultivate positive affect or optimism? Predicting improvements in medical adherence following a positive psychology intervention in patients with acute coronary syndrome. Gen Hosp Psychiatry. 2019 Nov-Dec;61:125-129. doi: 10.1016/j.genhosppsych.2019.06.001. Epub 2019 Jun 4. PMID 31280918
- [Derived] Celano CM, Albanese AM, Millstein RA, Mastromauro CA, Chung WJ, Campbell KA, Legler SR, Park ER, Healy BC, Collins LM, Januzzi JL, Huffman JC. Optimizing a Positive Psychology Intervention to Promote Health Behaviors After an Acute Coronary Syndrome: The Positive Emotions After Acute Coronary Events III (PEACE-III) Randomized Factorial Trial. Psychosom Med. 2018 Jul/Aug;80(6):526-534. doi: 10.1097/PSY.0000000000000584. PMID 29624523